CLINICAL TRIAL: NCT01153815
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Chinese Subjects With Post-stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112958
Record Dates: First submitted 2010-06-17; First posted 2010-06-30 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-01

CONDITIONS: Cerebrovascular Accident
Keywords: efficacy; Spasticity, Post-Stroke; safety; Botulinum toxin type A; placebo; spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Sodium chloride
  Interventions: Drug: placebo
- GSK1358820(Botulinum Toxin Type A) (Experimental): GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox")
  Interventions: Drug: GSK1358820(Botulinum toxin type A)

INTERVENTIONS:
Drug: GSK1358820(Botulinum toxin type A) — GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox")
  Other Names: OnabotulinumtoxinA; Botox
  Arms: GSK1358820(Botulinum Toxin Type A)
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This trial is a multicenter, double-blind, randomized, placebo-controlled study to compare GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox") with placebo on the efficacy and safety of treatment in poststroke subjects with focal wrist, finger and in some cases, thumb spasticity. Approximately 168 subjects will be enrolled. Subjects will receive a single treatment session of intramuscular GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox") '200U or 240U (if thumb spasticity is present)' or placebo in a randomization ratio of 1:1. The subjects will be observed until 12 weeks post injection. Outcome measures include changes from baseline at every post injection visit as measured on the Modified Ashworth Scale (MAS), Disability Assessment Scale (DAS) and Global Assessment Scale. The primary efficacy endpoint is the change from baseline at week 6 for wrist flexor muscle tone as measured on the Modified Ashworth Scale. Safety parameters will also be measured including adverse events, vital signs (pulse and blood pressure) and clinical laboratory tests (haematology, serum chemistry and urinanalysis).

DETAILED DESCRIPTION:
The primary objective of this study is to confirm the superior efficacy of a single treatment session with GSK1358820 (Botulinum Toxin Type A, aslo known as "OnabotulinumtoxinA" or "Botox") '200U or 240U (if thumb spasticity is present)' over placebo in subjects with post-stroke upper limb spasticity of both wrist and fingers flexors as measured on the Modified Ashworth Scale (MAS).

This trial is a multicenter, double-blind, randomized, placebo-controlled, parallel group study comparing GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox") to placebo for the treatment of subjects with focal wrist, finger and in some cases, thumb spasticity post-stroke. Approximately 168 subjects will be enrolled. Subjects will receive a single treatment session with intramuscular injections of GSK1358820 (Botulinum Toxin Type A, also known as "OnabotulinumtoxinA" or "Botox") '200U or 240U (if thumb spasticity is present)' or placebo in a randomization ration of 1:1. The subjects will be observed until 12 weeks post injection.

Each completed subject will attend 7 clinic visits. The maximum study duration is 13 weeks per subject. The study includes a 1 week pretreatment period, during which the screening visit (visit 1) is to take place. Only one upper limb (meeting inclusion/exclusion criteria) will be evaluated and treated in the study. Subjects will receive a single intramuscular treatment with either investigated drug or placebo at day 0 (visit 2). There will be five post-injection follow-up visits at weeks 1, 4, 6, 8 and 12 (visits 3 to 7). Week 6 (visit 5) is designated as the primary visit for determining efficacy.

The primary endpoint is the change from baseline at week 6 for wrist flexor muscle tone as measured on the Modified Ashworth Scale (MAS). The secondary endpoints include The secondary endpoints include the area under curve (AUC) for the MAS wrist score change from baseline, change from baseline for wrist/finger/thumb flexor muscle tone as measured on MAS, Disability Assessment Scale and Global Assessment Scale. The safety measures include adverse events, clinical laboratory tests and pulse, blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

1. Subjects with upper limb spasticity who are at least 6 months post stroke and present with spasticity of both the wrist and fingers in the study limb.
2. Wrist flexor muscle tone of 3 or greater and finger flexor muscle tone of 2 or greater as measured on MAS (0 to 4).
3. At least one functional disability item (i.e., hygiene, dressing, pain, or cosmesis) with a rating of 2 or greater on DAS (0 to 3).
4. If using oral anti-spasticity medications, must be stable for at least 1 month prior to study enrolment
5. If using physical therapy, must be stable for at least 1 month prior to study enrolment.
6. Male or female 18 to 75 years old at the time of informed consent.
7. >=40kg in weight.
8. QTc criteria: (either QTcb or QTcf, machine or manual overread, males or females); include the following details as appropriate: QTc<450 millisecond (msec) or <480msec for subjects with Bundle Branch Block-values based on either single electrocardiogram (ECG) values or triplicate ECG averaged QTc values obtained over a brief recording period.
9. Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2xULN; alkaline phosphatase and bilirubin ≤1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
10. In the opinion of the investigator, subject must clearly understand the intent of the study and be willing and able to comply with study instructions and complete the entire study.
11. Informed consent has been obtained.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Presence of fixed contracture of the study limb (absence of passive range of motion).
2. Profound atrophy of muscles to be injected (in the investigators opinion).
3. Infection or dermatological condition at the injection sites.
4. Significant inflammation in the study limb limiting joint movement.
5. History of or planned treatment for spasticity with phenol or alcohol block in the study limb.
6. History of or planned surgical intervention for spasticity of the study limb.
7. History (within 3 months of qualification) of or planned (during study period) casting of the study limb.
8. Participation in another clinical study currently, or within the 30 days immediately prior to enrolment.
9. Previous or current botulinum toxin therapy of any serotype.
10. Planned or anticipated initiation of new antispasticity medications during the clinical study.
11. Any medical condition that may put the subject at increased risk with exposure to GSK1358820, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might have interfered with neuromuscular function.
12. Concurrent use of aminoglycoside antibiotics or other agents that might interfere with neuromuscular function. A full list of prohibited medications that interfere with neuromuscular transmission is provided as Appendix 1.
13. Current treatment for spasticity with an intrathecal baclofen.
14. Females who are pregnant, nursing, or planning a pregnancy during the study period, or females of childbearing potential, not using a reliable means of contraception.
15. Known allergy or sensitivity to study medication or its components.
16. Bedridden subjects.
17. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
18. Presence of clinically unstable severe cardiovascular, renal or respiratory disease.
19. Investigator's opinion that the subject has a concurrent condition(s) that may put the subject at significant risk, may confound the study results, or may interfere significantly with the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Haerbin, Heilongjiang
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo 4 milliliters (mL) was injected into the wrist and finger muscles. 0.8 mL was injected into the thumb muscles if thumb spasticity was present during the 12-week study (once at Week 0).
- BTX 200 U: Botulinum Toxin Type A (BTX or GSK1358820) 200 Units (U) (4 mL) was injected into the wrist and finger muscles. 40 U (0.8 mL) was injected into the thumb muscles if thumb spasticity was present during the 12-week study (once at Week 0).
Period: Overall Study
Arm/Group | Placebo | BTX 200 U
Started | 83 | 87
Completed | 74 | 82
Not Completed | 9 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BTX 200 U | Total
Number analyzed (Participants) | 83 | 87 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (12.23) | 55.4 (10.69) | 55.8 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 65 | 64 | 129
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 83 | 87 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 6 for Wrist Flexor Muscle Tone as Measured on the Modified Ashworth Scale (MAS)
Description: The investigator, physiotherapist, or occupational therapist extended the participant's wrist as quickly as possible to grade flexor muscle tone. The MAS wrist score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at Week 6 was calculated as the value at Week 6 minus the value at Baseline.
Time Frame: Baseline (Day 0) and Week 6
Population: Full Analysis Set (FAS) Population: all randomized and treated participants. The missing data imputation method was used for analysis. For each participant, missing data points were replaced by the mean of the non-missing scores from both treatment groups for that variable at the specific visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale | -0.56 (0.735) | -1.21 (0.936)
Statistical Analysis 1: Comparison: Placebo vs BTX 200 U; Test type: Superiority or Other; p < 0.001, Exact Smirnov test

2. Secondary Outcome: Area Under the Curve (AUC) for the Change From Baseline at Weeks 6 and 12 for MAS Wrist Score
Description: The MAS wrist score was assessed by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Mean change from Baseline for the MAS wrist score was calculated as the value at Week 6 and Week 12 minus the value at Baseline. In a graph plotting time points on the horizontal axis (HA) and changes from Baseline on the vertical axis, the area surrounded by the MAS wrist score change curve and the HA was calculated and used as a summary index (AUC) for assessment of the MAS wrist score.
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 6 | -2.341 (2.8894) | -5.672 (4.3340)
  Week 12 | -5.618 (6.5412) | -12.712 (9.0510)

3. Secondary Outcome: Change From Baseline at Weeks 1, 4, 8, and 12 for Wrist Flexor Muscle Tone as Measured on the MAS
Description: The investigator, physiotherapist, or occupational therapist extended the participant's wrist as quickly as possible to grade flexor muscle tone. The MAS wrist score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at the indicated time points was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline (Day 0) and Weeks 1, 4, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 1 | -0.31 (0.504) | -0.80 (0.752)
  Week 4 | -0.46 (0.581) | -1.14 (0.843)
  Week 8 | -0.59 (0.757) | -1.27 (0.926)
  Week 12 | -0.48 (0.640) | -1.01 (0.822)

4. Secondary Outcome: Number of Participants Classified as Wrist Treatment Responders at All Post-injection Visits
Description: Wrist treatment responders were defined as participants with a decrease in wrist flexor muscle tone of at least one point on the MAS. The MAS wrist score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension).
Time Frame: Weeks 1, 4, 6, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
participants
  Week 1 | 24 | 51
  Week 4 | 33 | 63
  Week 6 | 36 | 62
  Week 8 | 36 | 64
  Week 12 | 23 | 54

5. Secondary Outcome: Change From Baseline at Weeks 1, 4, 6, 8, and 12 for Finger Flexor Muscle Tone as Measured on the MAS
Description: The investigator, physiotherapist, or occupational therapist extended the participant's finger as quickly as possible to grade the flexor muscle tone. The MAS finger score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at the indicated time points was calculated as the value at Week 1, 4, 6, 8, and 12 minus the value at Baseline.
Time Frame: Baseline (Day 0) and Weeks 1, 4, 6, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 1 | -0.30 (0.552) | -0.67 (0.769)
  Week 4 | -0.37 (0.654) | -0.98 (0.848)
  Week 6 | -0.42 (0.718) | -1.05 (0.879)
  Week 8 | -0.45 (0.683) | -1.04 (0.834)
  Week 12 | -0.28 (0.639) | -0.73 (0.773)

6. Secondary Outcome: Change From Baseline at Weeks 1, 4, 6, 8 and 12 for Thumb Flexor Muscle Tone as Measured on the MAS
Description: The investigator, physotherapist, or occupational therapist extended the participant's thumb as quickly as possible to grade the flexor muscle tone. The MAS thumb score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at the indicated time points was calculated as the value at Week 1, 4, 6, 8, and 12 minus the value at Baseline.
Time Frame: Baseline (Day 0) and Weeks 1, 4, 6, 8, and 12
Population: FAS Population. Only participants with thumb spasticity who received injection in the thumb muscles were evaluated. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 66 | 57
scores on a scale
  Week 1 | -0.33 (0.546) | -0.85 (0.841)
  Week 4 | -0.44 (0.655) | -1.02 (0.820)
  Week 6 | -0.53 (0.758) | -1.06 (0.844)
  Week 8 | -0.51 (0.804) | -1.06 (0.861)
  Week 12 | -0.43 (0.759) | -0.80 (0.797)

7. Secondary Outcome: Change From Baseline at Weeks 1, 4, 6, 8, and 12 for Principal Measure as Assessed on the Disability Assessment Scale (DAS)
Description: The investigator assessed 4 areas of disability, hygiene, pain, dressing, and limb posture, using the 4-point DAS (0=No functional disability to 3=Severe disability). Prior to the first dose, the investigator, in consultation with the participant, selected 1functional disability item (which had to have a score of 2 or greater as measured on the DAS, indicating moderate to severe disability) from the 4 areas of disability and assessed it as a principal measure. Change from Baseline at the indicated time points was calculated as the value at Weeks 1, 4, 6, 8, and 12 minus the value at Baseline.
Time Frame: Baseline (Day 0) and Weeks 1, 4, 6, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 1 | -0.13 (0.406) | -0.32 (0.560)
  Week 4 | -0.18 (0.446) | -0.49 (0.663)
  Week 6 | -0.28 (0.548) | -0.54 (0.696)
  Week 8 | -0.29 (0.594) | -0.59 (0.708)
  Week 12 | -0.29 (0.571) | -0.53 (0.676)

8. Secondary Outcome: Global Assessment Scale (GAS) Score as Evaluated by the Physician at the Indicated Time Points
Description: The physician used the GAS to assess response to treatment at each visit after injection. The assessor was the same throughout the study period. GAS scores were assessed by using the 9-point GAS (-4, -3, -2, -1, -0, +1, +2, +3, +4; -4=very marked worsenig, -0=unchanged, +4=very marked improvement) at the indicated time points.
Time Frame: Weeks 1, 4, 6, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 1 | 0.5 (0.80) | 1.2 (1.01)
  Week 4 | 0.7 (0.94) | 1.5 (1.08)
  Week 6 | 0.7 (1.04) | 1.5 (1.12)
  Week 8 | 0.7 (0.98) | 1.4 (1.08)
  Week 12 | 0.6 (0.86) | 1.2 (1.06)

9. Secondary Outcome: GAS Score as Evaluated by the Care Giver or the Participants at the Indicated Time Points
Description: The care giver or participants used the GAS to assess response to treatment at each visit after injection. The assessor was the same throughout the study period. GAS scores were assessed by using the 9-point GAS (-4, -3, -2, -1, -0, +1, +2, +3, +4; -4=very marked worsening, -0=unchanged, +4=very marked improvement) at the indicated time point.
Time Frame: Weeks 1, 4, 6, 8, and 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BTX 200 U
Number analyzed (Participants) | 83 | 87
scores on a scale
  Week 1 | 0.6 (0.81) | 1.1 (1.05)
  Week 4 | 0.7 (0.93) | 1.4 (1.14)
  Week 6 | 0.7 (1.06) | 1.5 (1.13)
  Week 8 | 0.7 (0.99) | 1.5 (1.08)
  Week 12 | 0.5 (0.85) | 1.2 (1.02)

ADVERSE EVENTS:
Arm/Group | Placebo | BTX 200 U
Serious Adverse Events (participants affected / at risk) | 1/83 | 2/87
Other Adverse Events (participants affected / at risk) | 21/83 | 16/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | BTX 200 U (N=87)
Cerebral infarction (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | BTX 200 U (N=87)
Blood bilirubin increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Lipids abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 2 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 2 | 0
Platelet count abnormal (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Bruxism (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.